CLINICAL TRIAL: NCT03346564
Title: Effects of a Ritual Training Program in the Head and Neck Cancer Patients: A Randomized Controlled Trial
Brief Title: Ritual Training Program in HNC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Shu-Ching Chen, Professor, Ministry of Science and Technology, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOST 103-2629-B-255 -001
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Education; Cognitive Change
Keywords: Head and neck cancer; Ritual training; disfigurement; body image
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ritual training program (Experimental): ritual training program for 8 weeks, biweekly
  Interventions: Behavioral: Ritual training program
- Routine care (Placebo Comparator): Routine care following hospital
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Ritual training program — Ritual training program including education and demonstration
  Arms: Ritual training program
Behavioral: Routine care
  Other Names: Routine care following hospital care
  Arms: Routine care

SUMMARY:
To evaluate the effects of a ritual training program in head and neck cancer (HNC) patients.

DETAILED DESCRIPTION:
The purpose of this study will to evaluate the effects of a ritual training program on disfigurement, self-esteem, social interaction, and body image in head and neck cancer (HNC) patients.

A prospective, repeated measures, randomized controlled therapeutic intervention design was employed. The experimental group will receive a ritual training program, and the control group will receive routine care. Patients will be assessed at three time points: baseline assessment (T0), and then at 1, 2, and 3-months (T1, T2, and T3) after participating in the ritual training program or routine care.

ELIGIBILITY:
Inclusion Criteria:

* > 20 years old,
* newly diagnosed first occurrence of HNC,
* completion of treatment and more than 3 months post-treatment

Exclusion Criteria:

* recurrence

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Disfigurement | Change from Baseline Disfigurement at 6 months
  Observer-rated disfigurement scale (1-9, higher score indicating greater levels of self-esteem higher disfigurement)
Body Image | Change from Baseline Body Image at 6 months
  Body Image Scale (0-30, higher scores indicate greater symptoms or distress in terms of body image concerns)
Social Interaction | Change from Baseline Social Interaction at 6 months
  Liebowitz Social Anxiety Scale(0-72, higher scores indicate greater fear or avoidance social interaction
Depression | Change from Baseline Depression at 6 months
  Hospital Anxiety and Depression Scale-Depression Subscale (0-21, higher score indicates a higher level of depression).
Self-Esteem | Change from Baseline Self-Esteem at 6 months
  Rosenberg Self-Esteem Scale(10-40, higher scores indicating greater levels of self-esteem)

IPD SHARING:
Plan to Share IPD: Undecided